CLINICAL TRIAL: NCT01401387
Title: Exocrine Pancreatic Insufficiency in Pancreatic Cancer: Evaluating the Need and Efficacy of Pancreatic Enzyme Replacement Therapy
Brief Title: Pancreatic Enzyme Suppletion in Pancreatic Cancer
Acronym: EPC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study never started
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPC 11-01; 2011-003373-28 (EudraCT Number)
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Pancreas; Normal Pancreatic Exocrine Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Active Comparator): Treatment with pancreatic enzymes after clinical sings and symptoms of steatorrhea and 10% decrease of weight at time of randomisation.
  Interventions: Other: Timing of start treatment with pancreatic enzymes
- Preventive treatment (Active Comparator): Patients will be prescribed with pancreatic enzymes immediately after diagnosis with pancreatic cancer, regardless of the presence of steatorrhea
  Interventions: Other: Timing of start treatment with pancreatic enzymes

INTERVENTIONS:
Other: Timing of start treatment with pancreatic enzymes — Patients who are randomised to standard treatment will start taking pancreatic enzymes only if they develop steatorrhea-related symptoms in combination with at least a 10% decrease in body weight (index weight at the time of randomisation).
  Other Names: Panzytrat 'HL'
  Arms: Standard treatment
Other: Timing of start treatment with pancreatic enzymes — Patients who are allocated to the anticipative group will start enzyme suppletion immediately and receive dietary consultation after randomization, regardless of symptoms.
  Other Names: Panzytrat 'HL'
  Arms: Preventive treatment

SUMMARY:
This study will evaluate the effect of immediate pancreatic enzyme suppletion on the physical and mental health status and survival of patients who are diagnosed with pancreatic cancer and are highly likely to develop exocrine pancreatic insufficiency during their disease process.

DETAILED DESCRIPTION:
Weight loss in cancer is caused by primary tumour effects and secondary effects (e.g. side effects of treatment, mechanical and intestinal obstruction). In pancreatic cancer, additional weight loss and malnutrition may be due to the development of exocrine pancreatic insufficiency (EPI). The presence of EPI in pancreatic cancer is frequently overlooked, because the focus of treatment is directed at possible surgery or chemotherapy and its potential side effects. Although studies have proven that pancreatic enzymes may prevent or decrease weight loss, they are seldom being prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the pancreas (histologically confirmed)
* Normal exocrine pancreatic function (Fecal Elastase test > 0.2 mg/g)
* Capable and willing to follow instructions given by the physician.

Exclusion Criteria:

* Other causes of fat malabsorption (celiac disease, IBD, and major gastrointestinal surgery).
* < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate if prescribing pancreatic enzymes in patients with pancreatic cancer leads to a decrease in weight loss. | every month during 6 months after inclusion
  Percentage of change in body weight ((index weight - monthly weight)/ index weight) x100% during the 6 months of follow-up. This will be measured on a monthly basis and measured by area under the ROC (Receiver Operating Characteristic) curve

SECONDARY OUTCOMES:
improvement of the nutritional status | every three months
  Nutritional deficiencies, 1 sample of blood will be drawn (3 times 8ml of blood):
  * Glucose, HbA1c (glycol Hb)
  * Magnesium, phosphate, ferritin
  * Hb
  * albumin
  * total protein
  * calcium
  * folic acid
  * vitamin A, E, B12
  * 1,25-di-OH-Vitamine D
  * 25-hydroxy vitamin D (25-OH-vitamin D)
quality-of-life | on a monthly base during 6 months after inclusion
  SF36 questionnaire
improvement of the nutritional status | every month during six months after inclusion
  A monthly patient journal which will focus on the presence or absence of steatorrhea-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- See also: Bruno MJ, Haverkort EB, Tijssen GP, Tytgat GN, van Leeuwen DJ. Placebo controlled trial of enteric coated pancreatin microsphere treatment in patients with unresectable cancer of the pancreatic head region. Gut. 1998 Jan;42(1):92-6. — http://www.ncbi.nlm.nih.gov/pubmed/9505892